CLINICAL TRIAL: NCT02941042
Title: This Trial is Conducted in the United State of America. The Aim of This Trial is to Investigate Safety, Tolerability and Pharmacokinetics for Single Doses of NNC9204-1177 in Subjects Being Overweight or With Obesity
Brief Title: A First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics for Single Doses of NNC9204-1177 in Subjects Being Overweight or With Obesity.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9277-4258; U1111-1173-8190 (Other: WHO)
Record Dates: First submitted 2016-10-07; First posted 2016-10-21 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC9204-1177 (Experimental)
  Interventions: Drug: NNC9204-1177
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC9204-1177 — A single dose administered subcutaneously ( s.c. under the skin)
  Arms: NNC9204-1177
Drug: Placebo — A single dose administered subcutaneously ( s.c. under the skin)
  Arms: Placebo

SUMMARY:
Trial Investigating Safety, Tolerability and Pharmacokinetics for Single Doses of NNC9204-1177 in Subjects being Overweight or with Obesity

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive) at screening

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol
* Subjects, aged at least 40 years, with an estimated 10-year atherosclerotic cardiovascular disease (ASCVD) (as described in the American College of Cardiology and the American Heart Association Prevention Guideline) risk above or equal to 5%
* Male subjects who are not sexually abstinent or surgically sterilised (vasectomy) and are sexually active with female partner(s) who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From time of dosing (day 1) until completion of the follow-up visit (day 39)

SECONDARY OUTCOMES:
Area under the NNC9204-1177 serum concentration-time curve | From 0 to 168 hours after a single s.c. dose
Maximum serum concentration of NNC9204-1177 | From time of dosing (day 1) until completion of the follow-up visit (day 39)
  Sampling was done day 1, 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 39
Time to maximum serum concentration of NNC9204-1177 | From time of dosing (day 1) until completion of the follow-up visit (day 39)
  Sampling was done day 1, 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 39
Change in body weight | Day 1, day 39
Change in QT interval corrected using the Fridericia formula (QTcF) | Day 1, day 39

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com